CLINICAL TRIAL: NCT06219980
Title: A Phase II Study of SBRT Followed by Neoadjuvant Chemoimmunotherapy of Sindilizumab Plus Docetaxel and Cisplatin for Locoregionally Advanced Squamous Carcinoma of Oral Cavity and Oropharynx
Brief Title: SBRT Followed by Neoadjuvant Chemoimmunotherapy of Sindilizumab Plus Docetaxel and Cisplatin for Locoregionally Advanced Squamous Carcinoma of Oral Cavity and Oropharynx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-278-01
Record Dates: First submitted 2024-01-04; First posted 2024-01-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: SBRT
Keywords: SBRT; immunotherapy; oral cancer; oropharyngeal cancer
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Combination Product: SBRT+chemoimmunotherapy

INTERVENTIONS:
Combination Product: SBRT+chemoimmunotherapy — All eligible patients will receive SBRT (6Gy*3 fractions, qod) to the primary site and metastatic lymph nodes. One week later, neoadjuvant chemoimmunotherapy of Sindilizumab (200mg) plus docetaxel (75mg/m2) and cisplatin (75mg/m2) will be administered every three weeks for three cycles. Then radical surgical resection will be performed and postoperative radiotherapy with or without chemotherapy will be supplemented according to the initial tumor staging and postoperative pathologic characteristics.

SUMMARY:
In resectable locally advanced oral cavity cancer and oropharyngeal cancer, SBRT with the total dose of 18 Gy by three fractions will be delivered to the primary tumor and metastatic lymph nodes every other day. One week later, neoadjuvant chemoimmunotherapy of Sindilizumab (200mg) plus docetaxel (75mg/m2) and cisplatin (75mg/m2) will be administered every three weeks for three cycles. Then radical surgical resection will be performed and postoperative radiotherapy with or without chemotherapy will be supplemented according to the initial tumor staging and postoperative pathologic characteristics. The investigators aim to evaluate the pathological complete response rate and safety of the combined treatment of SBRT with chemoimmunotherapy in locally advanced cancers of oral cavity and oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed squamous carcinoma of oral cavity or oropharynx
* III-IVa based on the eighth edition of AJCC
* aged 18 to 70
* ECOG PS 0-1
* no organ dysfunction
* Expected survival ≥ 3 months

Exclusion Criteria:

* diagnosed with other malignant tumors
* has autoimmune diseases or serious mental illness
* at high risk of hemorrhage
* Systemic or local glucocorticoid therapy within 4 weeks
* Comorbidities requiring long-term treatment with immunosuppressive drugs or systemic or topical corticosteroids in immunosuppressive doses
* Patients with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to screening.
* Prior use of anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, or anti-CTLA-4 antibody
* HIV or HCV
* HBsAg positive with positive HBV DNA copy number (quantitative test) ≥1000cps/ml

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
rate of pathological complete response | immediately after the surgery
  pathological complete response rate after radical resection

SECONDARY OUTCOMES:
rate of major pathological response | immediately after the surgery
objective response rate | two weeks after the chemoimmunotherapy
disease free survival | 3-year
overall survival | 3-year
rate of adverse events | one month after the postoperative radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darragh LB, Knitz MM, Hu J, Clambey ET, Backus J, Dumit A, Samedi V, Bubak A, Greene C, Waxweiler T, Mehrotra S, Bhatia S, Gadwa J, Bickett T, Piper M, Fakhoury K, Liu A, Petit J, Bowles D, Thaker A, Atiyeh K, Goddard J, Hoyer R, Van Bokhoven A, Jordan K, Jimeno A, D'Alessandro A, Raben D, McDermott JD, Karam SD. A phase I/Ib trial and biological correlate analysis of neoadjuvant SBRT with single-dose durvalumab in HPV-unrelated locally advanced HNSCC. Nat Cancer. 2022 Nov;3(11):1300-1317. doi: 10.1038/s43018-022-00450-6. Epub 2022 Nov 25. PMID 36434392
- [Background] Ma TM, Wong DJ, Chai-Ho W, Mendelsohn A, St John M, Abemayor E, Chhetri D, Sajed D, Dang A, Chu FI, Xiang M, Savjanji R, Weidhaas J, Steinberg ML, Cao M, Kishan AU, Chin RK. High Recurrence for HPV-Positive Oropharyngeal Cancer With Neoadjuvant Radiation Therapy to Gross Disease Plus Immunotherapy: Analysis From a Prospective Phase Ib/II Clinical Trial. Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):348-354. doi: 10.1016/j.ijrobp.2023.04.029. Epub 2023 May 2. No abstract available. PMID 37141981